CLINICAL TRIAL: NCT05441072
Title: Validation of Bulbicam for Use on Patient Suffering From Diabetic Retinopathy (DR) and Age-related Macular Degeneration (AMD)
Brief Title: Validation of Bulbicam for DR- and AMD-patients
Status: Completed | Type: Observational
Sponsor: Meddoc (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Prof Stig Larsen, Professor, Meddoc
Other Study IDs: V1-OTH /DR; AMD-I/2022
Record Dates: First submitted 2022-06-16; First posted 2022-07-01 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Retinopathy; Age-Related Macular Degeneration
MeSH Terms: conditions — Diabetic Retinopathy; Macular Degeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Diabetic Retinopathy (DR): Patients suffering from DR of both genders above 18 years of age with different disease degree. Each patient will be measured with BulbiCam device 6 times within three days
  Interventions: Device: BulbiCam
- Healthy controls DR: Gender- and age-matched healthy controls without any eye disease to the DR patients
  Interventions: Device: BulbiCam
- Age related macular degeneration (AMD): Patients suffering from AMD of both genders above 18 years of age with different disease degree.
  Interventions: Device: BulbiCam
- Healthy controls AMD: Gender- and age-matched healthy controls without any eye disease to the AMD patients
  Interventions: Device: BulbiCam

INTERVENTIONS:
Device: BulbiCam — The multi-test device, BulbiCam (BCAM), is a combined eye tracking; pupil metric; video graphic dual device which include the following 10 tests under development and ready for validation:
  1. 26 grids glaucoma screening perimetry
  2. 64 grids full perimetry (NeuroField64)
  3. Pupil and Relative Afferent Pupil Defect (RAPD) assessment
  4. Semi-automatic ptosis (droopy eyelid) grading
  5. Video-based nystagmus test
  6. Dynamic acuity and contrast sensitivity test
  7. Dark adaptation test
  8. Smooth pursuit eye movements
  9. Saccade movements
  10. Eye fixation stability
  BCAM is connected to the BulbiHub software where measured data is stored and presented in numbers, diagrams, and graphs.

SUMMARY:
Aim

* To investigate repeatability and stability of the six OTH-related Bulbicam tests in patients suffering from a) Diabetic retinopathy (DR), b) Age related macular degeneration (AMD) and matched healthy controls (HC).
* To compare Bulbicam and the Standard Method on measurements of Visual Field and Pupil
* To contribute to the establishment of normal range for DR and AMD patients with different degree in the disease development related to the Bulbicam tests.
* To contribute to the establishment of normal range for a normal population without eye-disease related to the Bulbicam tests. Study population The study consists of the following three study populations: 1) Patients suffering from DR of both genders above 18 years of age with different disease degree; 2) Patients suffering from AMD of both genders above 18 years of age with different disease degree; 3) Gender- and age-matched HC without any eye diseases.

Study procedure Participants, who fulfil the inclusion criteria; do not meet any of the exclusion criteria and willing to give informed consent to participate will receive an appointment for starting the study. The Bulbicam examination will be performed twice a day with a rest period of one hour between each registration. This procedure will be repeated the following two days. All demographic data, social factors and history of disease will be recorded at screening. Additionally, the quality of life (QoL) questionnaires EQ-5D-5L developed by EuroQol will be recorded initially as individual baseline values.

The Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be used for measuring and classifying the tolerability and toxicity at the end of each day of investigation.

DETAILED DESCRIPTION:
Aim

* To investigate repeatability and stability of the six OTH-related Bulbicam tests in patients suffering from a) Diabetic retinopathy (DR), b) Age related macular degeneration (AMD) and matched healthy controls (HC).
* To compare Bulbicam and the Standard Method on measurements of Visual Field and Pupil
* To contribute to the establishment of normal range for DR and AMD patients with different degree in the disease development related to the Bulbicam tests.
* To contribute to the establishment of normal range for a normal population without eye-disease related to the Bulbicam tests. Study population The study consists of the following three study populations: 1) Patients suffering from DR of both genders above 18 years of age with different disease degree; 2) Patients suffering from AMD of both genders above 18 years of age with different disease degree; 3) Gender- and age-matched HC without any eye diseases.

Trial equipment Bulbicam will be used in the study and the following six tests will be performed at each investigation: "Neurofield 64", "Ptosis", "Dynamic Acuity", "Dynamic Contrast ", "Dark Adaptation" and "Pupil RAPD". The Standard Method will be used initially for measurements of "Neurofield64", "Visual Field" and "pupil".

Design

The study will be performed as a controlled, open, and non-randomized, stratified observational multicenter study. The stratification factors are the pathology of DR and AMD and the degree of disease. Within each of the four strata, healthy matched controls related to gender- and age (1:1) will be included. The degree of DR is defined as follows:

1. Mild retinopathy: Mild nonproliferative diabetic retinopathy
2. Moderate retinopathy: Moderate nonproliferative diabetic retinopathy

The degree of AMD is defined as follows:

1. Early AMD
2. Intermediate For each included patient, a gender- and age-matched HC will be included. All included participants will perform Bulbicam eye-investigation twice at three flowing days with a rest period of at least one hour. Each investigation includes same six Bulbicam tests. The Standard method will only be performed once as the first investigation at day 1 for measurements of "Visual Field" and Pupil"

Variables The main variables will be the variables recorded at the six Bulbicam tests The supporting variables will be recorded by the Standard (ST) investigation for DR and AMD.

The central variables related to DR and AMD will be "RAPD NDF", "Seen /unseen "," Time until the given point is recorded as seen", "the light in decibel when the point is seen", X- and Y-coordinates and "Pupil diameter in mm" and "OCT RNFL ".

Study procedure Participants, who fulfil the inclusion criteria; do not meet any of the exclusion criteria and willing to give informed consent to participate will receive an appointment for starting the study. The Bulbicam examination will be performed twice a day with a rest period of one hour between each registration. This procedure will be repeated the following two days. All demographic data, social factors and history of disease will be recorded at screening. Additionally, the quality of life (QoL) questionnaires EQ-5D-5L developed by EuroQol will be recorded initially as individual baseline values.

The Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be used for measuring and classifying the tolerability and toxicity at the end of each day of investigation.

Sample size Sixteen DR patients and 16 AMD patients from each of the two categories will be recruited from the two participating hospitals. All together a total of 16x2=32 patients will be included. For each included patient, one gender- and age-matched HC will be recruited. In total 32 HC.

ELIGIBILITY:
Inclusion Criteria:

* Consists of patients diagnosed with either DR or AMD of both gender; passed the age of 18 years without any other eye disease; suffering from other know serious disease.

but have a health situation in accordance with expectations related to the age.

* Gender- and age-matched controls to patients in study population 1 or 2; passed the age of 18 years without any eye diseases; not suffering from other know serious disease and have a health situation in accordance with expectations related to the age.

Exclusion Criteria:

* Other visual disturbances and blindness
* Posterior Chamber Intra Ocular Lens (PCIOL)
* Physical or psychiatric disease, which may disturb the measuring procedure
* Patients who are not able to perform eye movements, so no full paresis of any ocular muscles.
* Patients whose visual acuity is less more than 1 logMAR in any eye, as these will not be able to focus on the test stimuli.
* Patients whose visible part of the eye is abnormal, such as subconjunctival hemorrhages or deformed pupils.
* Patients whose pupils are not able to respond normally to dilation or contraction due to damaged nerves, mechanical damage of the pupil etc.
* Participating in another clinical trial with pharmaceuticals the last six weeks before start of this trial treatment.
* With known alcoholic and drug dependency
* Not able to understand information.
* Not willing to give written consent to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of DR, AMD patients and healthy controls fulfilling the inclusion criteria and avoiding the exclusion criteria
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Visual Field | 0 hours
  Saccadic Reaction Time
Visual Field | 2 hours
  Saccadic Reaction Time
Visual Field | 4 hours
  Saccadic Reaction Time
Visual Field | 24 hours
  Saccadic Reaction Time
Visual Field | 26 hours
  Saccadic Reaction Time
Visual Field | 28 hours
  Saccadic Reaction Time
Ptosis | 0 hours
  Margin to reflex distanse
Ptosis | 2 hours
  Margin to reflex distanse
Ptosis | 4 hours
  Margin to reflex distanse
Ptosis | 24 hours
  Margin to reflex distanse
Ptosis | 26 hours
  Margin to reflex distanse
Ptosis | 28 hours
  Margin to reflex distanse

CONTACTS AND LOCATIONS:
Overall Officials: Goran Petrovski, PhD, Study Director — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/72/NCT05441072/Prot_ICF_000.pdf